CLINICAL TRIAL: NCT05965310
Title: Randomized Control Trial of the Impact of a Virtual Psychological Intervention on the Outcomes of ACLR
Brief Title: Anterior Cruciate Ligament Recovery With Virtual Psychological Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Thomas Lynch, Principle Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16012
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Depression; Anterior Cruciate Ligament Injuries; Mental Health Issue
MeSH Terms: conditions — Depression; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: This study is a parallel arm prospective randomized-controlled trial.
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Post-Operative Rehabilitation (No Intervention): No intervention, patients will receive the standard level of care.
- Virtual Psychological Intervention (Active Comparator): An asynchronous course of pre- and post-operative CBT modules (VPI) will be delivered to patients in Group A as an adjuvant treatment to standard-of-care rehabilitation.
  Interventions: Behavioral: Virtual Psychological Intervention: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Virtual Psychological Intervention: Cognitive Behavioral Therapy — An asynchronous course of pre- and post-operative CBT modules (VPI) will be delivered to patients in Group A as an adjuvant treatment to standard-of-care rehabilitation.
  Arms: Virtual Psychological Intervention

SUMMARY:
The goal of this parallel arm prospective randomized control trial study is to compare outcomes in Anterior Cruciate Ligament Reconstruction (ACLR) Surgery patients after exposure to a virtual psychological intervention (VPI) versus standard care. The main question the investigators are asking is if virtual administration of psychological CBT modules will be an accessible and convenient vehicle to improve ACLR outcomes. Participants will be placed either into a treatment group receiving virtual modules of cognitive behavioral therapy in addition to standard of care ACLR surgery or the control group receiving only the standard of care ACLR surgery. The investigators hypothesize that ACLR patients in the VPI cohort will have improved return to sport and post operative outcomes compared to controls.

DETAILED DESCRIPTION:
This study is a parallel arm prospective randomized-controlled trial. The expected duration of the study is two years. Participants will be placed either into a treatment group receiving virtual modules of cognitive behavioral therapy in addition to standard of care ACLR surgery or the control group receiving only the standard of care ACLR surgery. Trial eligibility criteria are as follows: patients over the age of 12 undergoing first time ACLR with a HFH Sports Orthopedic surgeon. Eligible participants will be randomized using computerized random number generation into two groups: Group A and Group B. Both groups will receive the same standard post-operative rehabilitation protocol. An asynchronous course of pre- and post-operative CBT modules (VPI) will be delivered to patients in Group A as an adjuvant treatment to standard-of-care rehabilitation. Each session is designed to provide patients with different CBT strategies to augment their recovery. Sessions will be delivered virtually by trained health professionals. Participants in Group B will receive standard-of-care rehabilitation only. Demographic information and additional protected health information will be handled securely in a securedatabase. Pre-operative PROMIS and PHQ-2 scores will be obtained for both groups via electronic medical record abstraction. Primary endpoints are as follows: Return to sport, defined as return to pre-injury involvement in the patient's respective sport at 3, 6, 12, and 24 months. Secondary outcomes are as follows: Patient-Reported Outcome Measurement Information System (PROMIS) scores, a validated patient reported outcome instrument, Patient Health Questionnaire-2 (PHQ-2) scores, a validated depression screening questionnaire, ACL-Return to Sport after Injury (ACL-RSI) scores, a validated scale to measure the psychological impact of returning to sport following ACLR3, Post-operative opioid usage and Utilization of additional counseling options (i.e., referral to behavioral health services)

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 12 with ACL injuries undergoing ACLR with a Henry Ford Sports Orthopedic Surgeon
* First time ACLR on the injured knee

Exclusion Criteria:

* Patients undergoing revision ACL surgery
* Concomitant posterior cruciate ligament injury of the involved knee
* Systemic or local infection pre-operatively
* Systemic administration of any type of corticosteroid or immunosuppressive agents within 30 days of surgery
* History of rheumatoid arthritis, inflammatory arthritis, or autoimmune diseases
* Pregnancy

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients who Return to Sport at time set-points | 3,6,12 and 24 months
  Comparing number of patients who Return to sport, defined as return to pre-injury involvement in the patient's respective sport at 3, 6, 12, and 24 months in each trial group.
Patient-Reported Outcome Measurement Information System (PROMIS) scores for Physical Function and Pain Interference | 3,6,12, and 24 months
  Comparing in each trial group, A validated patient reported outcome instrument where 50 is the average reference score of the patient population and the standard deviation is 10. For PROMIS measures, higher scores equals more of the concept being measured (e.g., more Pain Interference, more Physical Function). Thus a score of 60 is one standard deviation above the average referenced population. This could be a desirable or undesirable outcome, depending upon the concept being measured.
Patient Health Questionnaire-2 (PHQ-2) scores | 3,6,12, and 24 months
  Avalidated depression screening questionnaire with 3 points or more meaning a positive screen
ACL-Return to Sport after Injury (ACL-RSI) scores | 3,6,12 and 24 months
  A validated scale to measure the psychological impact of returning to sport following ACLR. There are three domains: risk appraisal, confidence, and emotions. A total score between 0 and 100 is calculated by adding and averaging the scores for each item. Greater psychological preparation is indicated by higher scores.

SECONDARY OUTCOMES:
Post-operative opioid usage | 0-24 months post-operatively
  the amount of usage of opioid medication post-operatively
Number of patients with Utilization of additional counseling options (i.e., referral to behavioral health services) | 0-24 months post-operatively
  Utilization of additional counseling options (i.e., referral to behavioral health services)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Sean Lynch, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT05965310/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT05965310/ICF_001.pdf